CLINICAL TRIAL: NCT02629003
Title: Evaluation of Radiation Dose for [11C]Cimbi-36
Brief Title: [11C]Cimbi-36 Dosimetry
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gitte Moos Knudsen (Other)
Responsible Party: Sponsor-Investigator, Gitte Moos Knudsen, Chair, Professor, MD, DMSc, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: H-15001910
Record Dates: First submitted 2015-12-07; First posted 2015-12-11 (Estimated); Last update posted 2019-03-26 (Actual); Status verified 2019-03

CONDITIONS: Healthy
Keywords: Positron Emission Tomography; Serotonin; 5-HT2A; Radioligand; Radiation dosimetry; Radiation dosage
MeSH Terms: interventions — Cimbi-36

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- [11C]Cimbi-36 (Active Comparator): [11C]Cimbi-36
  Maximum of 600 Mega Becquerel (MBq) or 1.5 micrograms, single dose intravenous (I.V.)
  Interventions: Drug: [11C]Cimbi-36
- [11C]Cimbi-36-5 (Active Comparator): [11C]Cimbi-36-5
  Maximum of 600 Mega Becquerel (MBq) or 1.5 micrograms, single dose intravenous (I.V.)
  Interventions: Drug: [11C]Cimbi-36-5

INTERVENTIONS:
Drug: [11C]Cimbi-36
  Arms: [11C]Cimbi-36
Drug: [11C]Cimbi-36-5
  Arms: [11C]Cimbi-36-5

SUMMARY:
The purpose of this study is to determine the dosimetry for the Positron Emission Tomography (PET) tracer [11C]Cimbi-36 in two different Carbon-11 labelling positions. This information will contribute to determining whether [11C]Cimbi-36 can be optimized by changing the C-11 labelling position.

DETAILED DESCRIPTION:
Healthy subjects wil undergo a whole-body Positron Emission Tomography (PET) scan with the Serotonin 2A Receptor (5-HT2A) radioligand [11C]Cimbi-36 or [11C]Cimbi-36-5 to determine the effective radiation dose and radiation dose for selected organs.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age
* Signed informed consent

Exclusion Criteria:

* Present or former neurological disease, severe somatic or psychiatric disease, or medication thet can interfere with the test results.
* Pregnancy at the time of the scan
* Breastfeeding
* Alcohol or substance abuse
* Exposure to radiation (>10 millisievert (mSv)) within the last year, or significant exposure at work
* Allergy to any of the substances in the Investigational medicinal product (IMP) formulation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2015-12; Primary Completion 2018-10-10 (Actual); Study Completion 2018-10-10 (Actual)

PRIMARY OUTCOMES:
Effective dose and absorbed dose for selected organs | 0 - 120 minutes
  Based on the Positron Emission Tomography (PET) scan Time activity curves (TACs) will be generated and used for calculating the radiation doses for selected organs and over all effective radiation dose.

SECONDARY OUTCOMES:
Measurement of radioactive metabolites in plasma | 0 - 120 minutes
  Venous blood samples will be used to measure radioactive metabolites and parent compound in the blood, using radio-High-performance liquid chromatography (HPLC). The parameters will be parent radioactivity and metabolite radioactivity as a fraction (unitless) of total radioactivity in plasma over time (unit = minutes).
Measurement of radioactivity in plasma and whole blood | 0 - 120 minutes
  Venous blood samples will be used to measure radioactivity in plasma and whole blood. The measurement will be given as a ratio (unitless) of plasma radioactivity relative to whole blood radioactivity over time (unit = minutes).

CONTACTS AND LOCATIONS:
Overall Officials: Gitte M Knudsen, MD, DMSc, Study Chair — Neurobiology Research Unit, Rigshospitalet
Locations (1):
- Neurobiology Research Unit, Rigshospitalet, Copenhagen, Denmark